CLINICAL TRIAL: NCT00592267
Title: A Screening Protocol for Children and Adolescents With Bipolar and Bipolar Spectrum Disorder
Brief Title: Screening Protocol for Children and Adolescents With Bipolar and Bipolar Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2001-P-001247
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Pediatric Bipolar Disorder
Keywords: pediatric; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The objective of this protocol is to establish a comprehensive screening process for the evaluation of eligibility for entry in a clinical trial program for children and adolescents with bipolar disorder.

DETAILED DESCRIPTION:
To address the urgent therapeutic needs of children and adolescents ages 4-17 with pediatric bipolar disorder, we have designed a series of clinical trials aimed at evaluating critical components of the treatment needs of this under-served and under-researched population. This approach will allow us to provide a full complement of clinical trials that will meet the most pressing needs of the bipolar children and adolescents and their families who are currently awaiting treatment.

Although these protocols have received prior IRB approval, potential participants present with a widely varied set of complaints not always discernable in a telephone screening interview. This state of affairs makes it very difficult to ask subjects to sign a specific clinical protocol without obtaining additional clinical information. Because of this we are proposing potential subjects to consent to undergo an in-depth clinical assessment that will allow subjects to be screened by a clinician for eligibility to a diverse clinical trials program available to them.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 4 to 17 inclusive with a suspected diagnosis of bipolar disorder.
* Subject and parent/ legal guardian must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their parent/ legal representative must be considered reliable.
* Each subject and his/her parent or authorized legal representative must understand the nature of the study. The subject's parent or authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
* One parent/ legal guardian must be able to accompany the subject to the clinic at each visit.

Exclusion Criteria:

* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Serious, unstable illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
* Mental retardation

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and Adolescents with symptoms of bipolar disorder
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-09; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Screening Protocol | Study Enrollment
  This protocol is a prescreening for other research studies.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Masschusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html